CLINICAL TRIAL: NCT06493084
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Dose Escalation Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LAE102 Injection in Healthy and Overweight/Obese Subjects
Brief Title: Evaluate LAE102 in Healthy and Overweight/Obese Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Laekna Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAE102CN1001
Record Dates: First submitted 2024-06-03; First posted 2024-07-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Overweight and Obese Volunteers
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part A LAE102 IV (Experimental): Single dose LAE102 by IV administration
  Interventions: Drug: LAE102 intravenous administration
- Part A placebo IV (Placebo Comparator): Single dose placebo by IV administration
  Interventions: Drug: placebo intravenous administration
- Part B LAE102 SC (Experimental): Single dose LAE102 by SC administration
  Interventions: Drug: LAE102 subcutaneous administration
- Part B placebo SC (Placebo Comparator): Single dose placebo by SC administration
  Interventions: Drug: placebo subcutaneous administration
- Part C LAE102 SC (Experimental): Multiple dose LAE102 by SC administration
  Interventions: Drug: LAE102 multiple subcutaneous administration
- Part C placebo SC (Placebo Comparator): Multiple dose placebo by SC administration
  Interventions: Drug: Placebo multiple subcutaneous administration

INTERVENTIONS:
Drug: LAE102 intravenous administration — A single dose of LAE102 administered intravenously
  Other Names: LAE102 IV
  Arms: Part A LAE102 IV
Drug: placebo intravenous administration — A single dose of placebo administered intravenously
  Other Names: Placebo IV
  Arms: Part A placebo IV
Drug: LAE102 subcutaneous administration — Single dose of LAE102 administered subcutaneously
  Other Names: LAE102 SC
  Arms: Part B LAE102 SC
Drug: placebo subcutaneous administration — single dose of placebo administered subcutaneously
  Other Names: Placebo SC
  Arms: Part B placebo SC
Drug: LAE102 multiple subcutaneous administration — Multiple dose of LAE102 administered subcutaneously
  Other Names: LAE102 SC
  Arms: Part C LAE102 SC
Drug: Placebo multiple subcutaneous administration — Multiple dose of placebo administered subcutaneously
  Other Names: Placebo SC
  Arms: Part C placebo SC

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of LAE102 injection in healthy and overweight/obese participants, and also evaluate the preliminary pharmacodynamic effect of multiple dose injections in overweight/obese participants.

DETAILED DESCRIPTION:
Part A is a randomized, double-blinded, placebo-controlled, single ascending dose by Intravenous (IV) administration in 40 Healthy participants;

Part B is a randomized, double-blinded, placebo-controlled, single ascending dose by subcutaneous (SC) administration in 24 Healthy participants;

Part C is a randomized, double-blind, placebo-controlled, multiple dose ascending and expanding by subcutaneous (SC) administration in 60 overweight/obese participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and aged 18 to 65 years (inclusive) at the screening visit
2. Male Body weight ≥ 50 kg, female Body weight ≥ 45 kg. For Part A&B, 18.5 ≤ BMI ≤ 28 kg/m². For part C, 26.0 ≤ BMI ≤ 40.0 kg/m²
3. Negative for human immunodeficiency virus antibody (HIV-Ab).
4. Female subjects with no childbearing potential or with childbearing potential which serum human chorionic gonadotropin (hCG) test must <5mIU/mL .
5. Male subjects are not allowed to donate sperm during this trial.
6. Voluntarily participate in the study and provide a signed and dated informed consent form.
7. Willing to comply with the scheduled visits, study treatment, laboratory tests, and other study-related procedures and requirements as stipulated in the study protocol.

Exclusion Criteria:

1. With clinically significant abnormalities in vital signs, physical examination, ECG or laboratory test results specified in the protocol.
2. Allergy to the investigational drug or its excipients, or a history of severe allergy (including any food or drug allergies).
3. Self-reported weight change is more than 5% in the previous 3 months prior to screening.
4. Diagnosed with secondary overweight or obesity.
5. Any clinically significant medical conditions and any diseases affecting the safety of the subject or the determination of study results.
6. History of major diseases or physical conditions in the central nervous system, respiratory system, cardiovascular system, digestive system, blood system, endocrine system, musculoskeletal diseases, mental illness, urinary system, or tumors, or any existing acute diseases, or other diseases or physical conditions that may affect the study or pose an unacceptable risk to the subjects.
7. Positive for hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV-Ab), or syphilis spirochete antibody (TP-Ab).
8. Known or suspected history of substance abuse or positive drug screening test.
9. Alcohol abuse within 1 year before screening or positive alcohol breath test at baseline.
10. Smoking more than 5 cigarettes per day within 3 months before screening, or unable to comply with the prohibition of smoking during the study period.
11. Received any vaccine within 30 days prior to screening, or planned to receive any vaccine during the study period.
12. Inability to ensure no use of any drugs, including prescription and non-prescription drugs (excluding paracetamol, ibuprofen, and topically applied eye/nasal drops and ointments with no systemic exposure risk), vitamins, supplements and herbal medicines, from 14 days before the initial administration (if the half-life of the drug used exceeds 14 days, then 5 half-lives shall apply) until the last visit period.
13. Participated in any clinical trial and received an investigational medicine or medical device within 3 months prior to dosing of the investigational product.
14. Underwent major surgery within 30 days before the initial administration or planned to undergo major surgery during the study period.
15. Donated blood or experienced blood loss ≥400 mL within 3 months before screening or received a blood transfusion.
16. Have special dietary requirements and cannot comply with a standardized diet.
17. History of fainting or syncope.
18. Dieting or receiving weight loss treatment within 30 days before the initial administration or experiencing major changes in lifestyle.
19. Use of GLP-1 receptor agonists, or weight loss medications or systemic corticosteroids (oral or intravenous for more than 7 days), or psychiatric medications within 3 months prior to the initial administration. Applicable to part C.
20. Regular engaged in muscle strength related exercise, applicable to part C.
21. Other situation that the investigator considers not appropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number & severity of participants with treatment-related adverse events as assessed by CTCAE V5.0 | From Day 1 to Day 29 for single dose part. From Day 1 to Day 196 for multiple dose part
  Findings on physical examination, ECG, vital signs, and reports of the laboratory results based on the CTCAE v5.0

SECONDARY OUTCOMES:
characterize the peak of serum concentration (Cmax) of LAE102 injection in healthy subjects | From pre-dose to Day 29 for single dose part. From pre-dose to Day 196 for multiple dose part.
  For both intravenously guttae & subcutaneous injection, to evaluate the maximum observed serum concentration(Cmax)
characterize the area under the serum concentration versus time curve (AUC) of LAE102 injection in healthy subjects | From pre-dose to Day 29 for single dose part. From pre-dose to Day 196 for multiple dose part.
  For both intravenously guttae & subcutaneous injection, to evaluate the area under the serum concentration versus time curve (AUC)
evaluate the expression levels of Activin A in blood samples | From pre-dose to Day 29 for single dose part. From pre-dose to Day 196 for multiple dose part.
  The validated methodology was employed to assay serum levels of Activin A in biological samples.
Incidence of positive Anti-drug antibody(ADA) after administration | pre-dose to Day 29 for single dose part. From pre-dose to Day 196 for multiple dose part.
  Test ADA status in biological sample via validated methodology

OTHER OUTCOMES:
Preliminary pharmacodynamic of total body weight for multiple dose part | From pre-dose to Day 168.
  Changes and percentage changes in total body weight (kg) after administration
Preliminary pharmacodynamic of lean mass for multiple dose part | From pre-dose to Day 168.
  Changes and percentage changes in lean mass after administration
Preliminary pharmacodynamic of fat mass for multiple dose part | From pre-dose to Day 168.
  Changes and percentage changes in fat mass after administration
Preliminary pharmacodynamic of thigh muscle volume for multiple dose part | From pre-dose to Day 168
  Changes and percentage changes in thigh muscle volume after administration
Preliminary pharmacodynamic of bone mineral density(BMD) for multiple dose part | From pre-dose to Day 168
  Changes and percentage changes in BMD after administration
BMI/waist circumference change and percentage. | From pre-dose to Day 29 forsingle dose. From pre-dose to Day 196 for multiple dose.
  Assess the Body Mass Index (BMI)/waist circumference change and percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Xuening Li, Professor, Principal Investigator — Zhongshan hospital affiliated to Fundan University
Locations (1):
- Fudan Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No